CLINICAL TRIAL: NCT04403893
Title: Feasibility and Safety of a Dedicated Biliary Stent for Transmural EUS-guided Hepatico-gastrostomy: the FIT Study
Acronym: FIT
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2753
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Malignant Bilio-pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: HANARO biliary stent placement — HANARO biliary stent placement

SUMMARY:
One of the major roles of interventional EUS is biliary drainage (EUS-BD) as an alternative to ERCP-based biliary decompression.

In fact, even when performed by expert endoscopists, ERCP-based stenting fails in 5% of cases. In these cases, standard alternative approaches include surgical bypass and percutaneous transhepatic cholangiography and biliary drainage (PTBD). However, these procedures are associated with higher patient discomfort and prolonged hospital stay.

The most diffuse approach for EUS-BD are choledochoduodenostomy (CDS) or hepaticogastrostomy (HGS). As a matter of fact, since dedicate devices as lumen apposing metal stents (LAMS), have been adopted for CDS, we have been witnessing the escalation of such procedure.

On the other hand, the diffusion of EUS-HGS is still limited due to the complexity of the procedure and the lack of dedicated devices. However, recently a dedicated stent was conceived as asymmetrically covered and shaped in order to have its uncovered, tubular end into the intrahepatic ducts and the covered, flanged end into the gastric cavity, to reduce the risk of migration. The developement of such stent could further increase both the technical feasibility and the clinical outcomes of HGS in order to explore the whole potential of this procedure and to definitively find its role in biliary drainage algorithm.

ELIGIBILITY:
Inclusion Criteria:

• subjects with malignant bilio-pancreatic diseases with an indication to undergo biliary stent positioning for biliary drainage after ERCP failure.

Exclusion Criteria:

* Age < 18 y
* Contra-indication for endoscopy or interventional radiology
* Unsigned informing consent form, ICF
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with malignant bilio-pancreatic diseases with an indication to undergo biliary stent positioning for biliary drainage after ERCP failure.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
AE and SAE events | 12 Months
  To assess the technical safety for EUS-guided hepaticogastrostomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No